CLINICAL TRIAL: NCT06879509
Title: The Use of Thromboelastography in Burn Injury to Improve Burn Coagulopathy Evaluation and Intervention
Brief Title: Thromboelastography to Study Burn Coagulopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Francesco Egro (Other)
Responsible Party: Sponsor-Investigator, Francesco Egro, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY23120009
Record Dates: First submitted 2024-12-06; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Burn; Coagulation, Blood
Keywords: burn; coagulation; Thromboelastography
MeSH Terms: conditions — Burns; Thrombosis | interventions — Thrombelastography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Burn Thromboelastography Group (Experimental): Overall study population (all participants are in the same group). See eligibility for further details.
  Interventions: Diagnostic Test: Thromboelastography

INTERVENTIONS:
Diagnostic Test: Thromboelastography — All participants will receive this intervention. Thromboelastography (TEG) is a blood test that provides a detailed assessment of the clotting process, measuring how blood clots form, strengthen, and dissolve. It offers real-time insights into a patient's coagulation status, helping to identify clotting disorders and guide treatment decisions.
  Other Names: TEG

SUMMARY:
This pilot study examines the use of thromboelastography (TEG), a specialized blood test, to evaluate clotting abnormalities in burn patients. The study aims to understand how burn injuries impact the body's ability to form and break down blood clots over time. Specifically, the investigators will research whether the percentage of total body surface area burned (%TBSA) is associated with changes in blood clotting, track the evolution of clotting patterns during the first four weeks following a burn injury, and explore whether these changes can predict recovery or complications. By providing new insights into clotting dynamics in burn patients, the study seeks to improve diagnostic methods, enhance monitoring strategies, and guide treatments to optimize patient care and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with acute burn injuries
* Aged 18 years and older
* Provided consent to participate in the study

Exclusion Criteria:

* Patients with a history of venous thromboembolism or hyper/hypocoagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Thromboelastography | Duration of hospital length of stay, up to 28 days
  Thromboelastography (TEG) evaluates blood's clotting ability by measuring the strength and elasticity of a clot over time, producing a dynamic graph. The following outcome measures will be assessed at specific time points (Day 1, Day 7, Day 14, Day 21, and Day 28):
  1. Reaction Time (R) (seconds) - The time from test initiation until the first detectable clot formation.
  2. Kinetic Time (K) (seconds) - The time from initial clot formation to a defined clot strength threshold.
  3. Maximum Amplitude (MA) (millimeters) - The peak strength of the formed clot.
  4. Alpha Angle (degrees) - The slope of the clot formation curve, representing the rate of clot development.
  5. Lysis at 30 Minutes (Ly30) (percentage of MA) - The percentage of clot degradation occurring 30 minutes after reaching maximum amplitude.
  Each parameter will be measured at the specified time points, and values will be aggregated into one TEG graph.

SECONDARY OUTCOMES:
Hospital Length of Stay | Duration of hospital length of stay, up to 28 days
  The investigators will measure the number of days patients stay in the hospital for treatment.
Complications During Treatment | Duration of hospital length of stay, up to 28 days
  The investigators will record any complications, such as infections, graft loss, flap loss, or thrombosis that occur during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco M Egro, MD, MSc, MRCS, Principal Investigator — Department of Plastic Surgery, University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared upon reasonable request by the peer-reviewed journal in which this study is published, provided the request is in alignment with ethical and legal standards.

REFERENCES:
- [Background] Baumeister S, Koller M, Dragu A, Germann G, Sauerbier M. Principles of microvascular reconstruction in burn and electrical burn injuries. Burns. 2005 Feb;31(1):92-8. doi: 10.1016/j.burns.2004.07.014. PMID 15639372
- [Background] Alessandri-Bonetti M, Kasmirski JA, Liu HY, Corcos AC, Ziembicki JA, Stofman GM, Egro FM. Impact of Microsurgical Reconstruction Timing on the Risk of Free Flap Loss in Acute Burns: Systematic Review and Meta-Analysis. Plast Reconstr Surg Glob Open. 2024 Aug 9;12(8):e6025. doi: 10.1097/GOX.0000000000006025. eCollection 2024 Aug. PMID 39129846